CLINICAL TRIAL: NCT00592150
Title: Effect of Gene Variants on Dopamine Receptor Natriuretic Responses (RMC033)
Brief Title: Effect of Gene Variants on Dopamine Receptor Natriuretic Responses
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert M. Carey, MD, Distinguished Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13072
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: Essential Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Fenoldopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Fenoldopam infusion
  Interventions: Drug: fenoldopam
- 2 (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fenoldopam — The fenoldopam infusion rate will be 0.05 μg/kg/min for 3 hours
  Arms: 1
Drug: Placebo — Placebo infusion for 3 hours
  Arms: 2

SUMMARY:
Hypothesis to be tested: Dopamine D1-like receptor-induced natriuresis is impaired in humans with G protein-related kinase 4 gene variants.

Our research group has discovered a D1 receptor/adenylyl cyclase coupling defect in renal PTCs from subjects with essential hypertension. We have found increased GRK-4 activity in renal PTCs in human essential hypertension due to activating variants of GRK-4, an effect that was reproduced in a transfected cell model. Preventing the translation of GRK-4 normalized the coupling of the D1 receptor to adenylyl cyclase in hypertension. Gene variants of GRK-4 cause a ligand-independent serine-phosphorylation of the D1 receptor, resulting in its uncoupling from the G-protein/effector complex. The desensitization of the D1 receptor in the renal PTC is hypothesized to be the cause of the compromised natriuretic effect of DA that eventually leads to Na+ retention and hypertension. The primary objective of this protocol is to demonstrate that natriuresis engendered by D1-like receptor activation with fenoldopam is blunted in subjects with 3 or more SNPs of GRK-4 compared with responses in subjects with 0-2 SNPs.

DETAILED DESCRIPTION:
Dopamine (DA) is an endogenous catecholamine, which serves as a biochemical precursor of norepinephrine and epinephrine. DA is well known as a neurotransmitter in the central nervous system. During the past decade, however, DA has been characterized as an important modulator of BP, Na+ balance, renal and adrenal function through an independent peripheral dopaminergic system. Evidence indicates that DA is synthesized locally within the kidney and acts at adjacent cells in an autocrine or paracrine fashion to control renal Na+ excretion (1,2).

The renin-angiotensin system (RAS) is a coordinated hormonal cascade, the principal effector of which is angiotensin II (ANG II). All of the components of the RAS are present within the kidney and intrarenal formation of ANG II provides major regulation of renal hemodynamic and tubule function via a self-contained intrarenal RAS (3,4). We propose to study the interaction of the renal dopaminergic and renin-angiotensin systems in the regulation of Na+ balance and Na+ sensitivity of blood pressure (BP) and in the pathophysiology of essential hypertension in man.

Our group has discovered a D1 receptor/adenylyl cyclase coupling defect in renal PTCs from subjects with essential hypertension. We have found increased GRK activity in renal PTCs in human essential hypertension due to activating variants of GRK-4, an effect that was reproduced in a transfected cell model. Preventing the translation of GRK-4 normalized the coupling of the D1 receptor to adenylyl cyclase in hypertension. The variants of GRK-4 cause a ligand-independent serine-phosphorylation of the D1 receptor, resulting in its uncoupling from the G-protein/effector complex. The desensitization of the D1 receptor in the renal PTC may be the cause of the compromised natriuretic effect of DA that eventually leads to Na+ retention and hypertension. Therefore, a primary objective of the entire Program Project Grant, of which this protocol is one part, is to identify humans with salt-sensitive hypertension and resistance to the inhibitory effect of D1-like receptor agonist fenoldopam on renal proximal Na+ reabsorption and determine whether these individuals have the activating polymorphisms of GRK-4 alone or in combination with polymorphisms of genes of the RAS.

Subjects are selected (on the basis of their GRK-4 genotype) from the pool of subjects that have already been genetically screened under IRB-HSR # 11494.

Subjects will be prepared and will be studied in approximate metabolic balance at 150 meq Na+/d. After approximate metabolic balance is achieved (estimated 5 days), subjects will receive either fenoldopam infusion or vehicle infusion on Day 6 and the opposite agent (fenoldopam or vehicle) will be infused on Day 7. The order of infusion will be randomized and the study will be conducted in double-blind fashion. Vehicle will be D5W and will be infused during the control period using the same rate as the post control period. At 1100 h on study Day 6, an i.v. infusion of fenoldopam or vehicle will be initiated and continued for 3h. The fenoldopam infusion rate will be 0.05 μg/kg/min. This infusion rate of fenoldopam has resulted in a greater than 2-fold increase in UNaV without alteration of systemic hemodynamic function in normal subjects (30). Plasma fenoldopam levels will be monitored to document delivery of this agent into the circulation. BP and heart rate will be measured in duplicate every 10 min during the experimental period (1100-1400h). The experimental period will be followed by a 2-hour post-control period (1400h-1600h) during which vehicle will be infused. Blood and urine samples will be obtained every 30 min and will be analyzed for Na+, K+, lithium and creatinine concentrations and osmolality. In addition, blood samples will be analyzed for PRA, cyclic AMP (blood and urine), plasma ANG II and aldosterone concentrations at 1045, 1215, 1345 and 1545 h. After completion of a post-control period at 1600h, the subjects will be allowed to be out of bed but remain as inpatients and receive the same diet as previously. No food is given after 2400h on Day 6. On Day 7, the identical protocol as on Day 6 will be repeated except that the opposite agent (fenoldopam or vehicle) will be infused. The subjects will be discharged from the GCRC on their previous diet.

ELIGIBILITY:
Inclusion Criteria:

Normotensive (NT) Subjects

* Men and women between ages of 18 and 70 years (inclusive)
* BMI of 18-29 (inclusive).
* Healthy as determined by updated full medical history, physical exam and:
* Standard 12-lead EKG
* Complete blood count and differential
* Fasting blood chemistry (metabolic screen and liver enzymes), lipid panel (cholesterol, triglycerides, HDL and LDL cholesterol)
* Urinalysis with microscopy.

Hypertensive (HT) Subjects

* Men and women between ages of 18 and 70 years (inclusive)
* BMI of 18-29 (inclusive).
* Mild to moderate hypertension
* Established by prior diagnosis
* Or established with screening (sitting) diastolic blood pressure in the range of 90 to 114 mm
* Healthy as determined by updated full medical history and physical exam and:
* Standard 12-lead EKG
* Complete blood count and differential
* Fasting blood chemistry (metabolic screen and liver enzymes), lipid panel (cholesterol, triglycerides, HDL and LDL cholesterol)
* Urinalysis with microscopy.

Exclusion Criteria:

* Younger than 18; 71 and older
* History of malignant or accelerated hypertension
* Contraindication to discontinuing anti-hypertensive medications
* Currently taking clonidine
* Impaired renal function (serum creatinine > 1.5 mg/dl) or urinary protein excretion > 200 mg/day or continuing active urinary sediment
* Myocardial infarction, cerebrovascular accident or transient ischemic attack
* Congestive heart failure by history and physical examination, severe peripheral vascular disease
* Glaucoma as determined by the referring physician
* Pregnancy or nursing
* Failure to give informed consent or comply with the protocol
* Systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 114 mm Hg (based on the mean of three consecutive measurements) following a three-week withdrawal of antihypertensive medications
* Protocol violations such as: failure to discontinue anti-hypertensive medications, failure to be admitted to the GCRC and complete failure to adhere to the prescribed diet.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Urine sodium excretion | 7 days

SECONDARY OUTCOMES:
gene dose effect of GPK-4 on fenoldopam induced natriuresis | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Carey, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States